CLINICAL TRIAL: NCT03638336
Title: Evaluation of the Performance of a Robotic Flexible Ureteroscopy (ILY) in Laser Treatment of Nephrolithiasis in the Upper Urinary Tract
Brief Title: Evaluation of the Performance of a Robotic Flexible Ureteroscopy (ILY) in Laser Treatment of Nephrolithiasis
Acronym: EASILY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No actual DM
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDIL/2016/SD-01
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Lithiasis, Urinary
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- flexible ureteroscopy (Experimental)
  Interventions: Device: ILY robotic flexible ureteroscopy

INTERVENTIONS:
Device: ILY robotic flexible ureteroscopy — fragmentation of nephrolithiasis

SUMMARY:
In this pilot study, we wish to evaluate the performance of a robotic flexible ureteorscopy (ILY) in the treatment of nephrolithiasis in the superior excretory system

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient has a single kidney stone in the calyx or the pelvis between 5 and 15mm something to do with a JJ probe
* Patient has an indication for in situ lithotripsy by supply ureteroscopy

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The patient is under safeguard of justice or state guardianship
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is pregnant or breastfeeding
* Patient treated with anticoagulants
* Documented untreated urinary infection within the previous 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of procedures performed entirely using the telemanipulator | end of study: 3 months
Number of procedures where the surgeon had to switch to manual mode or dedock the device | end of study: 3 months
If telemanipulator remained stable during procedure | end of procedure; less than 2 hours
  Yes/no
Time of procedure | end of procedure; less than 2 hours
Docking time | end of procedure; less than 2 hours
  time between docking of device and use of gamepad
Time taken to track kidney stones | end of procedure; less than 2 hours
Time taken for complete exploration of renal cavities | end of procedure; less than 2 hours
Laser fragmentation time | end of procedure; less than 2 hours
Speed of fragmentation | end of procedure; less than 2 hours
  mm3/minute
Any joint pain strain experienced by the surgeon before and after intervention | end of procedure; less than 2 hours
  binary yes/no
Satisfaction of surgeon in using the device | end of procedure; less than 2 hours
  Custom-made questionnaire with 3 sections measuring: ease of use, ergonomics in exploration of renal cavities and stability during fragmentation of laser

SECONDARY OUTCOMES:
Describe the rate of intra-operative complications during procedure | end of procedure; less than 2 hours
Describe the rate of intra-operative complications | 1 month
Integrity of the ureroscope at the end of the procedure | end of procedure; less than 2 hours
  binary yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Droupy, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No